CLINICAL TRIAL: NCT04692636
Title: Investigating the Impact of Blood Pressure Variability on the Outcomes of Hemodialysis Vascular Access
Brief Title: BP Variability on the Outcomes of Hemodialysis Vascular Access
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Other Study IDs: 106-033-E
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Hemodialysis Access Failure; Blood Pressure; Dialysis Access Malfunction
Keywords: hemodialysis access failure; blood pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total study cohort: Patients with dysfunctional hemodialysis vascular access referred for PTA or patients who received maintenance hemodialysis will be prospectively enrolled.
  Interventions: Diagnostic Test: Measure: BP measurements, inter-dialysis BP variability, intra-dialysis hypotension

INTERVENTIONS:
Diagnostic Test: Measure: BP measurements, inter-dialysis BP variability, intra-dialysis hypotension — BP will be measured at the beginning and end of each dialysis session in a seated position by a trained dialysis nurse in accordance with the routine unit practice and entered into an electronic database. BP was measured using validated oscillometric BP monitor equipped in hemodialysis machines (Fresenius 4008S or Nikisso DBB-05), which were maintained as per dialysis unit protocols.

SUMMARY:
Hemodialysis vascular access dysfunction continues to be a major source of morbidity and mortality in patients with ESRD. Thrombosis is the most common cause of secondary vascular access failure Although intimal hyperplasia at the outflow vein is the most common cause of thrombosis, 20-40% of thrombosis may develop secondary without underlying anatomic abnormalities. Low-flow states secondary to low BP have been proposed to precipitate access thrombosis. In previous studies, lower pre- and post- dialysis SBP are associated with a higher rate of access thrombosis. Nonetheless, high blood pressure is also a well-known risk factor for arteriosclerosis, intimal hyperplasia, and thrombotic vascular events. In dialysis patients, the relation between blood pressure and thrombosis seems to be more complex, and few studies have delineated the effect of blood pressure in a systematic manner.

In addition to the static component of blood pressure, blood pressure variability (BPV) is increasingly accepted as a novel risk factors for vascular disease. BPV is categorized as either long or short term. In dialysis patients, long-term BPV is typically defined on the basis of BP measurements taken at the start of hemodialysis (inter-dialysis BPV); short-term BPV is usually considered in terms of variability during hemodialysis (intra-dialysis BPV). BP variability is increased in ESRD patients and is associated with adverse outcomes. To the best of our knowledge, only one study by Cheung et al focused on intra-dialytic BPV, which found intradialytic hypotension to be a risk factor for access thrombosis. Nonetheless, access thrombotic events rarely occur during the dialysis session. It remained unclear that if inter-dialysis BPV is a more relevant factor for access thrombosis. Answer to this question is of clinical significance because the optimal BP target after PTA remained unknown. In this study, we aimed to investigate the effect of BP variability on the outcomes of hemodialysis vascular access, major cardiovascular events in maintenance hemodialysis patients. We also aimed to evaluate the determinants of BPV in hemodialysis patients, including medication, frailty, fluid status and autonomic function. The impact of autonomic function and frailty on the outcomes of vascular access and cardiovascular events will be evaluated as well.

DETAILED DESCRIPTION:
Hemodialysis vascular access dysfunction continues to be a major source of morbidity and mortality in patients with ESRD1. After the publication of the dialysis outcome quality initiative guidelines, endovascular interventions gradually replaced surgical revisions as the primary treatment of dysfunctional dialysis access2. Although percutaneous transluminal angioplasty (PTA) can achieve a high success rate, recurrent stenosis and thrombosis are usually inevitable3, 4. As a result, repeated interventions are required and cause a substantial financial burden on the health care system. Intimal hyperplasia at the outflow vein is the most common cause of vascular access dysfunction5. Thrombosis may develop secondary to outflow venous stenosis, but it can also develop without underlying anatomic abnormalities6.

Thrombosis is the most common cause of secondary vascular access failure (i.e., failure of functioning vascular access) and is associated with luminal stenosis in 60% to 80% of cases. However, because 20% to 40% of cases of access thrombosis occur in the absence of stenosis, and because not all stenotic accesses thrombose, other factors must contribute to access thrombosis.7 Among other factors, low-flow states secondary to low BP have been proposed to precipitate access thrombosis.8 These putative causes of access thrombosis make intuitive sense, but few studies have actually examined these factors in a systematic manner.

The relation between blood pressure and access thrombosis is complex. Very few studies have addressed on this issue. Unlike in the general population, blood pressure is not linearly associated with adverse outcomes in hemodialysis patients. Traditionally, high blood pressure is a well-known risk factors of intimal hyperplasia and thrombosis. Nonetheless, lower BP may also lead to decreased access blood flow, which has been shown to independently predict subsequent access thrombosis.9 In addition to the static component of blood pressure, blood pressure variability (BPV) is closely associated with adverse outcomes in patients with or at risk of vascular disease than 'usual' BP.10 They may play a causal role in the progression of organ damage and in triggering vascular events. BPV is categorized as either long or short term, based on the time interval over which it is considered.11 Long term BPV is usually measured as visit-to-visit BPV and can be considered in intervals of days, weeks or months. In the dialysis patients, the long term BPV is typically defined on the basis of BP measurements taken at the start of hemodialysis treatment (inter-dialytic BPV). Short-term BPV is usually measured by ambulatory BP monitoring or during specified short-time intervals. Among dialysis patients, short-term BPV can be considered in terms of variability that occurred during hemodialysis treatment (intra-dialytic BPV).

4 BP variability is known to be increased in patients with ESRD.12 Among patients undergoing hemodialysis, potential causes of high BP variability such as baroreceptor dysfunction, aortic stiffness, and variations in intravascular volume, as well as plausible outcomes such as cerebral small-vessel disease, cerebral hemorrhage, and cardiac sudden death are increased compared to the general population.13, 14 Therefore, increased BP variability may provide a potential explanation for access thrombosis among patients undergoing hemodialysis. Currently, only one study by Cheung et al has focused on the effect of BP variability. Lower pre-and post- dialysis SBP is associated with a higher rate of access thrombosis, consistent with previous studies.15, 16 More importantly, intradialytic hypotension is also a risk factor for access thrombosis and may account for some of the 20% to 40% of cases without obvious structural abnormalities.16 Nonetheless, most access thrombotic events did not occur during the dialysis session. It remained unclear if inter-dialysis BP variability is also a risk factor for vascular access thrombosis. The answer to these queries is of therapeutic relevance because the achievement of the recommended target BP in dialysis patients may be associated with higher rates of inter- or intra-dialytic hypotension.17 Accordingly, we aimed to investigate the effect of intra-dialysis BPV, inter-dialysis BPV, and intra-dialysis hypotension on thrombosis of hemodialysis vascular access.We also aimed to evaluate the determinants of BPV in hemodialysis patients, including medication, frailty, fluid status and autonomic function. The impact of autonomic function and frailty on the outcomes of vascular access and cardiovascular events will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* age from 20-99 years old, undergoing regular hemodialysis for at least six months.

Exclusion Criteria:

* (1) patients received regular dialysis less than 6 months
* (2) patients with clinical evidence of acute or chronic inflammation, decompensated heart failure, recent myocardial infarction, or unstable angina in recent 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dysfunctional hemodialysis vascular access referred for PTA or patients who received maintenance hemodialysis will be prospectively enrolled.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular access thrombosis | 30 months
  An access that had clotted without blood flow

SECONDARY OUTCOMES:
Post-intervention primary patency | 30 months
  the time until next intervention on the access of any kind
Post-intervention secondary patency | 30 months
  time from enrollment until surgical revision or abandonment of the access
stroke (both ICH and infarction) | 5 years
  time from enrollment to the first event
major cardiovascular events | 5 years
  CV death, non-fatal MI, non-fatal stroke, and acute/critical limb ischemia

OTHER OUTCOMES:
impact of frailty on vascular access events | 30 months
  enrollment to the first vascular access events
impact of frailty on vascular access thrombosis | 30 months
  enrollment to the first vascular access thrombosis
impact of frailty on cardiovascular events | 5 years
  enrollment to the first cardiovascular events

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsinchu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsieh MY, Chuang SY, Lee CK, Luo CM, Cheng CH, Liao MT, Lin PL, Yang TF, Wu CC. Risks and outcomes of critical limb ischemia in hemodialysis patients: a prospective cohort study. Clin Kidney J. 2022 Dec 8;16(3):585-595. doi: 10.1093/ckj/sfac263. eCollection 2023 Mar. PMID 36865012